CLINICAL TRIAL: NCT00188032
Title: Strategies for Suspected Pulmonary Embolism in Emergency Departments - SPEED Study
Brief Title: Strategies for Suspected Pulmonary Embolism in Emergency Departments
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Angers (Other Government)
Collaborators: Ministry of Health, France (Other Government)
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: PHRC-04-01
Record Dates: First submitted 2005-09-12; First posted 2005-09-16 (Estimated); Last update posted 2009-02-05 (Estimated); Status verified 2009-02

CONDITIONS: Quality of Health Care; Pulmonary Embolism
Keywords: pulmonary embolism; clinical practice; quality of health care; diagnostic criteria; Computer-Assisted Decision Support; reminders
MeSH Terms: conditions — Pulmonary Embolism

INTERVENTIONS:
Procedure: Computer-Assisted diagnostic Decision Support
Procedure: written diagnostic guidelines
Procedure: electronic therapeutic reminders

SUMMARY:
Aims: 1) To evaluate the effectiveness of two interventions aimed at improving the management of patients with suspected pulmonary embolism: Written guidelines and Computer-Assisted Decision Support (CADS). 2) To evaluate the impact of electronic reminders on the appropriateness of the treatment of patients with suspected PE

Design: Pragmatic, unblinded, cluster randomised controlled study.

Setting: 20 French Emergency Departments

Patients: Out patients suspected of having pulmonary embolism

Methods: Emergency physicians will prospectively complete a standardized electronic form on Personal Data Assistant (PDA), including patients' characteristics, the clinical probability if assessed, the diagnostic tests performed, the treatments initiated and the final diagnostic and therapeutic decisions. Patients will be interviewed at the end of a 3-month follow-up period using a standardized questionnaire.

The reference rate of appropriateness of the diagnostic management before intervention will be assessed in each centre. At the end of this preliminary period, the centres will be randomized in two fold two groups according to a factorial design with stratification on their reference level of appropriateness. Half of the centres will have written guidelines and half a Computer-Assisted Decision Support for the diagnosis of PE on the PDA. In each of these two main groups, half of the centres will have electronic reminders on their PDA concerning the treatment of PE.

Judgment criteria

Main : Rate of strategies considered as validated according to the results of the systematic review and meta-analysis.3

Secondary judgment criteria (diagnosis):

* Rate of strategies considered as validated or acceptable according to the opinion of international advisors.
* Rate of thromboembolic-events during a 3-month follow-up period in patients for whom pulmonary embolism will be ruled out
* Costs of the diagnostic management

Secondary judgment criteria (treatment):

* Delay between Emergency Department admission and the first dose of antithrombotic treatment in patients with high clinical probability of PE according to the Revised Geneva Score
* Rate of inappropriate treatment according to international recommendations for patients with confirmed PE.

Number of patients: By estimating that the rate of appropriateness would be 55% in the "written guidelines" group, 1331 patients are necessary to highlight an absolute superiority of 15% in the "CADS" group (rate of conformity of 70%).

The number of patients will be adjusted at the end of the preliminary period according to the level of appropriateness before interventions considering that it will improve less than 5% in the "written guidelines" group.

DETAILED DESCRIPTION:
Background: The management of patients with suspected pulmonary embolism (PE) represents an important medical and economic issue. In French Emergency Departments, more than 100 000 suspicions of PE are dealt with per year. In a previous work, we found that the routine diagnostic practice differs to a large extent from international guidelines and that excluding PE on the basis of inappropriate criteria exposes patients to a six-fold increased risk of venous thromboembolism during 3-months follow-up.1 Passive interventions to improve quality are generally ineffective but Computer-Assisted Decision Support and reminders appear as promising.2

Interventions:

At the end of the preliminary period, we will perform for all the investigators, an interactive oral presentation of the strategies considered as validated on the basis of a systematic review and meta-analysis.3 A strategy end up to exclude PE is considered as validated if the probability of PE is below 5% and a strategy end up to confirm PE is considered as validated if the probability of PE is upper than 85%. The strategies that do not achieve these criteria but considered as acceptable by international advisors will be presented too as well as the recommendations for the treatment of PE.4 In the group "written guidelines", emergency physicians will be provided with cards presenting the list of the validated and acceptable strategies as well as the Geneva diagnostic algorithm.5 The algorithm will be mention as a way to follow appropriate diagnostic criteria.

In the "CADS" group, the recommendations will be integrated into the electronic form allowing calculation of the pre-test probability according to revised Geneva Score 6, calculation of the post-test probabilities according to the likelihood ratios of the tests 3 and contextualized reminders as which test perform or when stop investigations.

In the groups "treatment help", reminders concerning the treatment (indications and contraindications, dosage) will be integrated into the electronic form on the PDA.

1. Roy PM, Meyer G, Vielle B, Legall C, Verschuren F, Furber A. Inappropriateness of Diagnostic Management in Patients with Suspected Pulmonary Embolism: Frequency, Predictors and Association with Outcome. J Thromb Haemost 2005; 3:OR 304.
2. Grimshaw JM, Shirran L, Thomas R, et al. Changing provider behavior: an overview of systematic reviews of interventions. Med Care 2001; 39:II2-45.
3. Roy PM, Colombet I, Durieux P, Chatellier G, Sors H, Meyer G. Systematic review and meta-analysis of strategies for the diagnosis of suspected pulmonary embolism. Bmj 2005; 331:259.
4. Buller HR, Agnelli G, Hull RD, Hyers TM, Prins MH, Raskob GE. Antithrombotic therapy for venous thromboembolic disease: the Seventh ACCP Conference on Antithrombotic and Thrombolytic Therapy. Chest 2004; 126:401S-428S.
5. Perrier A, Roy PM, Aujesky D, et al. Diagnosing pulmonary embolism in outpatients with clinical assessment, D-dimer measurement, venous ultrasound, and helical computed tomography: a multicenter management study. Am J Med 2004; 116:291-9.
6. Le Gal G, Righini M, Roy PM, et al. Derivation and validation of a simple standardized clinical score to predict pulmonary embolism in emergency patients: the revised geneva score. Ann Intern Med 2005; In press.

ELIGIBILITY:
Inclusion Criteria:

* patient with suspected pulmonary embolism
* prescription of a specific paraclinical diagnostic investigation or start of a specific treatment for pulmonary embolism

Exclusion Criteria:

* confirmation or exclusion of pulmonary embolism before admission in emergency department
* confirmation of deep venous thrombosis before admission in emergency department
* suspicion of pulmonary embolism during hospitalization (in-patient)
* suspicion of pulmonary embolism without investigation realization
* patient already included in the study
* patient refusing the utilization of his data for the study

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1331 (Estimated)
Dates: Start 2005-06; Study Completion 2006-09 (Actual)

PRIMARY OUTCOMES:
rate of agreement between the diagnostic criteria applied in daily practice and those validated in the scientific literature

SECONDARY OUTCOMES:
-(diagnostic intervention) Rate of strategies considered as validated or acceptable according to the opinion of international advisors.
- (diagnostic intervention) Rate of thromboembolic-events during a 3-month follow-up period in patients for whom pulmonary embolism will be ruled out
- (diagnostic intervention) Costs of the diagnostic management
- (therapeutic reminders) Delay between Emergency Department admission and the first dose of antithrombotic treatment in patients with high clinical probability of PE according to the Revised Geneva Score
- (therapeutic reminders)Rate of inappropriate treatment according to international recommendations for patients with confirmed PE.

CONTACTS AND LOCATIONS:
Overall Officials: Pierre-Marie Roy, MD, PhD, Principal Investigator — UH Angers
Locations (20):
- France (20):
  - H Argenteuil, Argenteuil
  - UH Besançon, Besançon
  - H Bethune, Béthune
  - UH Ambroise Pare, Boulogne-Billancourt
  - UH Caen, Caen
  - H Chalons en Champagne, Châlons-en-Champagne
  - H Chateauroux, Châteauroux
  - H Compiegne, Compiègne
  - UH Dijon, Dijon
  - H Dreux, Dreux
  - UH Grenoble, Grenoble
  - H Langres, Langres
  - H le Mans, Le Mans
  - H Lons le Saunier, Lons-le-Saunier
  - UH Nancy, Nancy
  - UH La Pitie Salpetriere, Paris
  - H Roanne, Roanne
  - H Saint Nazaire, Saint-Nazaire
  - H Thouars, Thouars
  - UH Toulouse, Toulouse

REFERENCES:
- [Background] Roy PM, Colombet I, Durieux P, Chatellier G, Sors H, Meyer G. Systematic review and meta-analysis of strategies for the diagnosis of suspected pulmonary embolism. BMJ. 2005 Jul 30;331(7511):259. doi: 10.1136/bmj.331.7511.259. PMID 16052017
- [Derived] Roy PM, Durieux P, Gillaizeau F, Legall C, Armand-Perroux A, Martino L, Hachelaf M, Dubart AE, Schmidt J, Cristiano M, Chretien JM, Perrier A, Meyer G. A computerized handheld decision-support system to improve pulmonary embolism diagnosis: a randomized trial. Ann Intern Med. 2009 Nov 17;151(10):677-86. doi: 10.7326/0003-4819-151-10-200911170-00003. PMID 19920268